CLINICAL TRIAL: NCT02514473
Title: A Phase 3, Double Blind, Placebo Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Lumacaftor in Combination With Ivacaftor in Subjects Aged 6 Through 11 Years With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Brief Title: A Study to Evaluate the Efficacy and Safety of Lumacaftor in Combination With Ivacaftor in Subjects With CF, Homozygous for the F508del-CFTR Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX14-809-109
Record Dates: First submitted 2015-07-23; First posted 2015-08-03 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LUM/IVA (Experimental): Fixed-dose combination with lumacaftor (LUM) 200 mg every 12 hours (q12h)/ ivacaftor (IVA) 250 mg q12h
  Interventions: Drug: VX-809; Drug: VX-770
- Placebo (Placebo Comparator): Matching placebo q12h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-809
  Other Names: lumacaftor
  Arms: LUM/IVA
Drug: Placebo
  Arms: Placebo
Drug: VX-770
  Other Names: ivacaftor
  Arms: LUM/IVA

SUMMARY:
To evaluate the efficacy and safety of lumacaftor in combination with ivacaftor in subjects aged 6 Through 11 years with cystic fibrosis (CF), homozygous for the F508del CF transmembrane conductance regulator (CFTR) mutation

ELIGIBILITY:
Inclusion Criteria:

* Subjects who weigh ≥15 kg without shoes a the Screening Visit
* Subjects with confirmed diagnosis of CF at the Screening Visit.
* Subjects who are homozygous for the F508del CFTR mutation
* Subjects with ppFEV1 of ≥70 percentage points adjusted for age, sex, and height
* Subjects with a screening LCI2.5 result greater than or equal to 7.5

Exclusion Criteria:

* History of any comorbidity reviewed at the Screening Visit that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Any clinically significant laboratory abnormalities at the Screening Visit that would interfere with the study assessments or pose an undue risk for the subject
* Clinically significant abnormalities in hemoglobin, liver function, or renal function at the Screening Visit.
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 28 days before Day 1
* History of solid organ or hematological transplantation at the Screening Visit

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (29):
  - Birmingham, Alabama
  - Los Angeles, California
  - Palo Alto, California
  - Aurora, Colorado
  - Wilmington, Delaware
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Omaha, Nebraska
  - Manchester, New Hampshire
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Salt Lake City, Utah
  - Colchester, Vermont
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (5):
  - Herston
  - New South Wales
  - Parkville
  - Subiaco
  - Westmead
- Belgium (2):
  - Brussels
  - Leuven
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec
- Copenhagen, Denmark
- France (3):
  - Bordeaux
  - Bron
  - Paris
- Germany (5):
  - Berlin
  - Cologne
  - Giessen
  - Hanover
  - Munich
- Stockholm, Sweden
- United Kingdom (4):
  - Edinburgh, Lothian Region
  - Leeds, West Yorkshire
  - Belfast
  - London

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Ratjen F, Hug C, Marigowda G, Tian S, Huang X, Stanojevic S, Milla CE, Robinson PD, Waltz D, Davies JC; VX14-809-109 investigator group. Efficacy and safety of lumacaftor and ivacaftor in patients aged 6-11 years with cystic fibrosis homozygous for F508del-CFTR: a randomised, placebo-controlled phase 3 trial. Lancet Respir Med. 2017 Jul;5(7):557-567. doi: 10.1016/S2213-2600(17)30215-1. Epub 2017 Jun 9. PMID 28606620

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 206 participants were randomized in the study, of which 204 participants were exposed to study treatment (101 participants received 'Placebo' and 103 participants received '(lumacaftor [LUM] / ivacaftor [IVA])'.
Groups:
- Placebo: Participants received placebo matched to LUM in combination with IVA fixed-dose combination (FDC) tablets orally every 12 hours (q12h) for 24 weeks.
- LUM/IVA: Participants received LUM 200 milligram (mg) in combination with IVA 250 mg FDC tablets orally q12h for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | LUM/IVA
Started | 101 | 103
Completed | 98 | 98
Not Completed | 3 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo matched to LUM in combination with IVA FDC tablets orally q12h for 24 weeks.
- LUM/IVA: Participants received LUM 200 mg in combination with IVA 250 mg FDC tablets orally q12h for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | LUM/IVA | Total
Number analyzed (Participants) | 101 | 103 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (1.59) | 8.7 (1.6) | 8.8 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 63 | 121
  Male | 43 | 40 | 83

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Lung Clearance Index 2.5 (LCI2.5) Through Week 24
Description: Lung clearance index (LCI) is a measure of ventilation inhomogeneity that is derived from a multiple breath washout test using Nitrogen (N2). LCI2.5 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value.
Time Frame: Baseline, Through Week 24
Population: Full Analysis Set (FAS) included all randomized participants who received any amount of study drug. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 99 | 99
Ratio | 0.08 (0.13) | -1.01 (0.13)
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Analysis was performed using mixed-effects model for repeated measures (MMRM). The model included treatment, visit and treatment-by-visit interaction as fixed effects; and participant as a random effect with adjustments for baseline, weight (less than [<] 25 kilogram [kg] versus greater than or equal to [>=] 25 kg) and percent predicted forced expiratory volume in 1 second (FEV1) severity (<90 versus >=90) at screening; Test type: Superiority; p < 0.0001, MMRM; Least Square (LS) Mean Difference = -1.09, 95% CI 2-sided [-1.43 to -0.75]

2. Secondary Outcome: Average Absolute Change From Baseline in Sweat Chloride at Day 15 and Week 4
Description: Sweat samples were collected using an approved collection device. Baseline was defined as the average of the measurements at screening and on Day 1 pre-dose. Change from Baseline in sweat chloride at Day 15 and Week 4 was calculated. The average of the 2 values (Change at Day 15 and Week 4) was reported.
Time Frame: Baseline, Day 15 and Week 4
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Millimole per liter (mmol/L)
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 94 | 95
Millimole per liter (mmol/L) | 0.8 (1.0) | -20.0 (1.0)

3. Secondary Outcome: Absolute Change From Baseline in Body Mass Index (BMI) at Week 24
Description: BMI was defined as weight in kg divided by height in square meter (m^2).
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Kg/m^2
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 97 | 98
Kg/m^2 | 0.27 (0.07) | 0.38 (0.07)

4. Secondary Outcome: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score Through Week 24
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Baseline, Through Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 78 | 76
Units on a scale | 3.0 (1.0) | 5.5 (1.0)

5. Secondary Outcome: Absolute Change From Baseline in Lung Clearance Index 5.0 (LCI5.0) Through Week 24
Description: LCI is a measure of ventilation inhomogeneity that is derived from a multiple breath washout test using Nitrogen (N2). LCI5.0 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/20th of its starting value.
Time Frame: Baseline, Through Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 99 | 99
Ratio | 0.08 (0.05) | -0.36 (0.05)

6. Secondary Outcome: Absolute Change From Baseline in Sweat Chloride at Week 24
Description: Sweat samples were collected using an approved collection device.
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 91 | 90
mmol/L | 3.2 (1.3) | -21.6 (1.3)

7. Secondary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) Through Week 24
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Wang standards were used to calculate ppFEV1 (for age, gender, race, and height).
Time Frame: Baseline, Through Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent predicted of FEV1
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 100 | 101
Percent predicted of FEV1 | -1.3 (0.8) | 1.1 (0.8)

8. Secondary Outcome: Relative Change From Baseline in ppFEV1 Through Week 24
Description: as for outcome 7
Time Frame: Baseline, Through Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 100 | 101
Percent change | -0.9 (1.0) | 2.2 (1.0)

9. Secondary Outcome: Absolute Change From Baseline in BMI-for-age Z-score at Week 24
Description: BMI was defined as weight in kg divided by height in m^2. z-score is a statistical measure to evaluate how a single data point compares to a standard. It describes whether a mean was above or below the standard. BMI, adjusted for age and sex, was analyzed as BMI-for-age z-score (BMI z-score). The BMI-for-age z-scores were calculated using National Center for Health Statistics growth charts.
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 97 | 98
Z-score | 0.05 (0.04) | 0.08 (0.04)

10. Secondary Outcome: Absolute Change From Baseline in Weight at Week 24
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Kg
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 97 | 98
Kg | 1.7 (0.2) | 2.0 (0.1)

11. Secondary Outcome: Absolute Change From Baseline in Weight-for-age Z-score at Week 24
Description: Z-score is a statistical measure to evaluate how a single data point compares to a standard. It describes whether a mean was above or below the standard. Weight, adjusted for age and sex, was analyzed as weight-for-age z-score (weight z-score). The weight-for-age z-scores were calculated using National Center for Health Statistics growth charts.
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 97 | 98
Z-score | 0.02 (0.02) | 0.06 (0.02)

12. Secondary Outcome: Absolute Change From Baseline in Height at Week 24
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Centimeter (cm)
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 97 | 98
Centimeter (cm) | 2.6 (0.1) | 2.9 (0.1)

13. Secondary Outcome: Absolute Change From Baseline in Height-for-age Z-score at Week 24
Description: Z-score is a statistical measure to evaluate how a single data point compares to a standard. It describes whether a mean was above or below the standard. Height, adjusted for age and sex, was analyzed as height-for-age z-score (height z-score). The height-for-age z-scores were calculated using National Center for Health Statistics growth charts.
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 97 | 98
Z-score | 0.00 (0.02) | 0.03 (0.02)

14. Secondary Outcome: Absolute Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) Domains Through Week 24
Description: The TSQM is a 14-item self-administered questionnaire which measures participants' experiences with their medication on four dimensions: effectiveness, side effects, convenience and global satisfaction. For each dimension, responses are added and transformed to a scale from 0 to 100, where higher scores indicate greater satisfaction.
Time Frame: Baseline, Through Week 24
Population: FAS. Here, 'Number of participants analyzed' = those participants who were evaluable for this endpoint and 'Number Analyzed' = those participants who were evaluable at the specified time points for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 91 | 91
Units on a scale
  Change Through Week 24: Effectiveness: number analyzed (Participants) | 91 | 90
  Change Through Week 24: Effectiveness | 0.6 (1.5) | 1.7 (1.5)
  Change Through Week 24: Side Effects: number analyzed (Participants) | 90 | 90
  Change Through Week 24: Side Effects | 0.4 (0.8) | -1.0 (0.8)
  Change Through Week 24: Convenience: number analyzed (Participants) | 90 | 91
  Change Through Week 24: Convenience | 9.9 (1.2) | 11.9 (1.2)
  Change Through Week 24: Global Score: number analyzed (Participants) | 90 | 90
  Change Through Week 24: Global Score | -2.3 (1.6) | -1.4 (1.6)

15. Secondary Outcome: Number of Pulmonary Exacerbation Events
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. The number of events were reported.
Time Frame: Baseline through Week 24
Population: FAS.
Measure: Number; unit: Pulmonary exacerbation events
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 101 | 103
Pulmonary exacerbation events | 18 | 24

16. Secondary Outcome: Percentage of Participants With At Least 1 Pulmonary Exacerbation Event
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms.
Time Frame: Baseline through Week 24
Population: FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 101 | 103
Percentage of participants | 14.9 | 19.4

17. Secondary Outcome: Time-to-first Pulmonary Exacerbation
Description: Time-to-first pulmonary exacerbation was analyzed using the Kaplan-Meier estimates. Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms.
Time Frame: Baseline through Week 24
Population: FAS.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 101 | 103
Days | NA [NA to NA] — Median and range was not reached as less than 50% of participants had the event of interest. | NA [NA to NA] — Median and range was not reached as less than 50% of participants had the event of interest.

18. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, inpatient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. Any AE that increased in severity or newly developed at or after initial dosing of study drug to Week 28 was considered treatment-emergent.
Time Frame: Baseline up to Week 28
Population: Safety Set included all participants who were exposed to any amount of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 101 | 103
participants
  Participants With Any Treatment-Emergent AEs | 98 | 98
  Participants With Treatment-Emergent SAEs | 11 | 13

19. Secondary Outcome: Average Pre-dose Concentration (Ctrough,Ave) and Average 3 to 6 Hours Post-dose Concentration (C3-6h,Ave) For Lumacaftor and Ivacaftor
Description: Ctrough,ave is average of individual pre-dose observed concentrations across Week 4 and 24. C3-6h,ave is average of individual 3 to 6 hours post-dose observed concentrations across Day 1, 15 and Week 4. This outcome was not planned to be assessed in Placebo arm.
Time Frame: For Ctrough,ave: before morning dose on Week 4 and 24; For C3-6h,ave: 3 to 6 hours after morning dose on Day 1, 15 and Week 4
Population: Pharmacokinetic (PK) set included all randomized participants who received any amount of study drug and had a PK assessment. Here, 'Number of participants analyzed' = those participants who were evaluable for this endpoint and 'Number Analyzed' = those participants who were evaluable at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | LUM/IVA
Number analyzed (Participants) | 102
Nanogram per milliliter (ng/mL)
  LUM: Ctrough,ave: number analyzed (Participants) | 99
  LUM: Ctrough,ave | 10200 (4460)
  LUM: C3-6h,ave | 20600 (6560)
  IVA: Ctrough,ave: number analyzed (Participants) | 99
  IVA: Ctrough,ave | 107 (91.2)
  IVA: C3-6h,ave | 821 (348)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 28
Arm/Group | Placebo | LUM/IVA
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/103
Serious Adverse Events (participants affected / at risk) | 11/101 | 13/103
Other Adverse Events (participants affected / at risk) | 98/101 | 98/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=101) | LUM/IVA (N=103)
Poor venous access (Vascular disorders) | 0 | 1
Procedural anxiety (Injury, poisoning and procedural complications) | 0 | 1
Bacterial test positive (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug interaction (General disorders) | 0 | 1
Device related thrombosis (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 2 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 5 | 8
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=101) | LUM/IVA (N=103)
Alanine aminotransferase increased (Investigations) | 8 | 8
Bacterial test positive (Investigations) | 8 | 7
Aspartate aminotransferase increased (Investigations) | 6 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 46
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 18
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 17
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 15
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Headache (Nervous system disorders) | 9 | 13
Pyrexia (General disorders) | 20 | 15
Fatigue (General disorders) | 11 | 9
Abdominal pain upper (Gastrointestinal disorders) | 7 | 13
Abdominal pain (Gastrointestinal disorders) | 10 | 10
Nausea (Gastrointestinal disorders) | 9 | 10
Vomiting (Gastrointestinal disorders) | 10 | 10
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 8 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 6
Decreased appetite (Metabolism and nutrition disorders) | 6 | 3
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 16 | 13
Upper respiratory tract infection (Infections and infestations) | 10 | 13
Rhinitis (Infections and infestations) | 5 | 6
Nasopharyngitis (Infections and infestations) | 8 | 5
Viral upper respiratory tract infection (Infections and infestations) | 8 | 5
Influenza (Infections and infestations) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: PI is free to publish results of the study after (1)first multi-center publication, (2)if sponsor elects not to publish the results, or (3)18 months after close of the study, whichever occurs first.Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.